CLINICAL TRIAL: NCT01514487
Title: A Randomised, Double-blind, Single-centre, Three-period, Cross-over Trial in Healthy Subjects Investigating the Bioequivalence Between Each of the Two New Liraglutide Formulations at pH 7.9 and 8.15 and the Planned Phase 3 Formulation at pH 7.7
Brief Title: Comparison of Three Liraglutide Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1636
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- pH 7.7 (Experimental)
  Interventions: Drug: liraglutide
- pH 7.9 (Experimental)
  Interventions: Drug: liraglutide
- pH 8.15 (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — One single dose of 0.75 mg administered on three different dosing occasions with a 14-day wash-out period between each dosing. Injected subtaneously

SUMMARY:
This trial is conducted in Oceania. The aim of this trial is to test for bioequivalence between each of the two new liraglutide formulations at pH 7.9 and 8.15 and the planned Phase 3 formulation at pH 7.7.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Good general health as judged by the investigator, based on medical history, physical examination including 12-lead ECG (electrocardiogram), vital signs and blood and urinary laboratory assessments.
* Body Mass Index (BMI) of 18-27 kg/m^2, both inclusive

Exclusion Criteria:

* History of any clinically significant renal, hepatic, cardiovascular, pulmonary, gastrointestinal,
* metabolic, endocrine, haematological, neurological, psychiatric disease or other major disorders
* that may interfere with the objectives of the study, as judged by the investigator
* Family or personal history of Primary hyperparathyroidism or pheochromocytoma or thyroid malignancy or multiple endocrine neoplasia
* Impaired renal function
* Uncontrolled treated/untreated hypertension
* Any clinically significant abnormal ECG
* Active hepatitis B and/or active hepatitis C
* Positive HIV (human immunideficiency virus) antibodies
* Known or suspected allergy to trial product(s) or related products
* Pregnant, breast-feeding or the intention of becoming pregnant or not using adequate contraceptive measures
* Prescription or non-prescription medication, except for paracetamol and vitamins
* History of alcoholism or drug abuse during the last 12 months
* Smoking of more than 10 cigarettes per day, or the equivalent for other tobacco products
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, soft drinks such as cola, chocolate) as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01-13 (Actual); Primary Completion 2005-03-30 (Actual); Study Completion 2005-03-30 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (0-t)
Cmax, maximum concentration

SECONDARY OUTCOMES:
Area under the curve (0-infinity)
tmax, time to reach Cmax
t½, terminal half-life
Terminal elimination rate constant
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Adelaide, Australia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com